CLINICAL TRIAL: NCT03772392
Title: Enhanced Recovery After Surgery for Hepatobiliary-Pancreatic Surgery
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18185
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2019-01

CONDITIONS: Liver Diseases; Pancreas Disease
MeSH Terms: conditions — Liver Diseases; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: HPB resection — :Liver and Pancreas surgery - Compliance with ERAS protocol

SUMMARY:
ERAS protocols have been utilized extensively in abdominal and non abdominal surgery over the past 20 years. These protocols incorporate evidence based, multi-disciplinary peri-operative care components. Compliance with these protocols is associated with reduced length of stay, reduced morbidity and reduced hospital costs.

ERAS protocols within HPB units are les well established with less evidence supporting their use. Liver resection protocols are increasing in use, but ERAS post Whipples resection is less established.

In the HPB unit at the Royal Infirmary of Edinburgh, the liver HPB protocol is in use but a recent audit identified that that the compliance rate is low with compliance rates as low as 30 per cent in some care domains.

DETAILED DESCRIPTION:
1.1 Background

Enhanced Recovery After Surgery(ERAS) protocols have been utilized extensively in abdominal and non abdominal surgery over the past 20 years. These protocols incorporate evidence based, multi-disciplinary peri-operative care components. Compliance with these protocols is associated with reduced length of stay, reduced morbidity and reduced hospital costs.

ERAS protocols within hepatobiliary pancreatic (HPB) units are les well established with less evidence supporting their use. Liver resection protocols are increasing in use, but ERAS post Whipples resection is less established.

1.2 RATIONALE FOR STUDY

In the HPB unit at the Royal Infirmary of Edinburgh, the liver HPB protocol is in use but a recent audit identified that that the compliance rate is low with compliance rates as low as 30 per cent in some care domains.

2. OBJECTIVES

To compare the compliance of ERAS protocol care components within an HPB unit before and after an education programme.

3. STUDY POPULATION

3.1 NUMBER OF PARTICIPANTS An attempt to observe 100 patients will be made over the study period. A preliminary audit of 27 patients has been performed.

4. PARICIPANT SELECTION

4.1 IDENTIFYING PARTICIPANTS

Those patients to be included will be identified from the theatre schedule as listed for HPB resectional surgery. Their compliance with the ERAS protocol will then be observed over the course of their stay.

4.2 CONSENT The ERAS protocol is part of the unit policy and so patients will not be undergoing any intervention that is not already part of normal practice and consent. Therefore further or additional consent will not be required.

5. DATA COLLECTION Over a six month period the compliance to the ERAS protocol will be assessed in patients undergoing HPB resections.

Compliance programme

1. Patients will be given an information leaflet describing their post-operative care pathway
2. Nursing and medical staff will receive education regarding the ERAS protocol and achievements
3. Auditing of the ERAS protocol adherence will subsequently be performed

Outcome measures

1. Functional recovery
2. Morbidity
3. Compliance rate of the individual peri-operative care components
4. Drop out rate
5. Length of stay
6. STATISTICAL ANALYSIS Chi squared analysis of dichotomised data will be performed. T test and Mann Whitney U tests will be performed to assess differences between the pre and post education programme results.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing open HPB resectional surgery within the HPB unit at the Royal Infirmary of Edinburgh

Exclusion Criteria:

* Laparoscopic surgery Non resectional surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Those patients to be included will be identified from the theatre schedule as listed for HPB resectional surgery. Their compliance with the ERAS protocol will then be observed over the course of their stay.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Time of functional recovery from surgery | 90 days
  Time to achieve discharge criteria post-operatively

SECONDARY OUTCOMES:
Morbidity | 90 days
  Post operative complications
Compliance | 90 days
  Adherence rates to ERAS protocol and individual ERAS components
Length of Stay | 90 days
  Time in hospital after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided